## **Clinical Trial Protocol**

**Protocol Title:** Multicenter, Randomized, Controlled, Double-Masked

> Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease (The

ONSET Study)

**Protocol Number:** OPP-002

**Study Phase:** 2

**Product Name:** OC-01 Nasal Spray

Dry Eye Disease **Indication: Investigators:** Multi-Center

Oyster Point Pharma, Inc. **Sponsor:** 

700 Alexander Park

Suite 301

Princeton, NJ 08540

**Contract Research Organization:** 

**Institutional Review** 

Board:



| | Date |
|--------------------|----------------|
| Original Protocol: | April 24, 2018 |
| Amendment 1: | July 11, 2018 |

#### **Confidentiality Statement**

This protocol contains confidential, proprietary information of and/or Oyster Point Pharma, Inc. Further dissemination, distribution or copying of this protocol or its contents is strictly prohibited.

#### **SPONSOR PERSONNEL**



### **MEDICAL MONITOR**




# **SYNOPSIS**

| Protocol Title: Protocol Number: Investigational Product: | A Multicenter, Randomized, Controlled, Double-Masked Clinical Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Signs and Symptoms of Dry Eye Disease OPP-002 OC-01 (varenicline tartrate) nasal spray: 0.02% (low dose), 0.1% (medium dose), and 0.2% (high dose) |
|---|---|
| Study Objective: | The objective of this study is to evaluate the safety and effectiveness of OC-01 Nasal Spray as compared to placebo on signs and symptoms of dry eye disease (DED) |
| | Overall Study Design |
| Structure: A Phase 2, multicenter, randomized, controlled, double masked study | |
| Duration: | Five study visits over approximately four weeks |
| Control: | Placebo (OC-01 Vehicle Nasal Spray) |
| Dosing Regimen: | Intranasal delivery of OC-01 twice daily (BID) for 4 weeks |
| Summary of Visit<br>Schedule: | <ul> <li>Visit 1 = Day 1, Screening and Treatment (Schirmer's Test Evaluation)</li> <li>Visit 2 = 7 ± 2, Treatment (Schirmer's Test Evaluation)</li> <li>Visit 3 = 14 ± 2, Treatment (Schirmer's Test Evaluation)</li> <li>Visit 4 = 21 ± 2, Treatment (Eye Dryness Score Evaluation)</li> <li>Visit 5 = 28 ± 2, Treatment (Schirmer's Test Evaluation)</li> </ul> |
| Measures Taken to Reduce Bias: | This is a randomized, double-masked study |
| Stu | udy Population Characteristics |
| Number of Subjects: | Approximately 160 (40 per arm) |
| Condition/Disease: | Dry Eye Disease |








# **Exclusion Criteria:** Subjects must not: 6. Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery (e.g. laser-assisted in-situ keratomileusis, laser epithelial keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1 10. Have a history or presence of any ocular disorder or condition in either eye that would, in the opinion of the Investigator, likely interfere with the interpretation of the study results or participant safety such as significant corneal or conjunctival scarring; pterygium or nodular pinguecula; current ocular infection, conjunctivitis, or inflammation not associated with dry eye; anterior (epithelial) basement membrane corneal dystrophy or other clinically significant corneal dystrophy or


degeneration; ocular herpetic infection; evidence of keratoconus; etc. Blepharitis not requiring treatment




| Sponsor: | Oyster | <b>Point</b> | Pharma, | Inc. |
|----------|--------|--------------|---------|------|
| | | | | - |

| Study Formulations: | Subjects will be randomized 1:1:1:1 to be treated with OC-01 nasal solution delivered as a 50 microliter (µL)-intranasal spray in each nostril at the following formulations: |
|---|---|
| | <ul> <li>0.02% OC-01 (varenicline tartrate) nasal spray [low dose]</li> <li>0.1% OC-01 (varenicline tartrate) nasal spray [medium dose]</li> <li>0.2% OC-01 (varenicline tartrate) [high dose]</li> <li>Placebo nasal spray (OC-01 Vehicle Nasal Spray)</li> </ul> |
| | Evaluation Criteria |
| Efficacy Measures: Primary Efficacy Measures: • Schirmer's Test at Visit 5 (Day 28) • Eye Dryness Score (EDS) at Visit 4 (Day 21) | |
| Safety Measures: | Adverse Event (AE) Query |
| Other Efficacy Measures: | <ul> <li>Patient-reported outcome: Ora Calibra® Ocular<br/>Discomfort Scale</li> <li>Corneal Staining</li> </ul> |
| Summary of Known and Potential Risks and Benefits to Human Subjects There are no known risks with the instillation of OC-01 (varenicline tartrate) nasal spray. | |


# **TABLE OF CONTENTS**

| Syno | psis | | 3 |
|---|---|---|---|
| Table | e of Co | ontents | 9 |
| List | of Abb | previations1 | 2 |
| 1 | Intro | duction1 | 3 |
| 2 | Study | Objectives1 | 4 |
| 3 | Clinic | eal Hypotheses1 | 4 |
| 4 | Overa | all Study Design1 | 5 |
| 5 | Study | Population1 | 5 |
| | 5.1 | Number of Subjects1 | 5 |
| | 5.2 | Study Population Characteristics1 | 5 |
| | 5.3 | Inclusion Criteria1 | 5 |
| | 5.4 | Exclusion Criteria1 | 6 |
| | 5.5 | Withdrawal Criteria1 | 8 |
| 6 | Study | Parameters1 | 8 |
| | 6.1 | Efficacy Measures1 | 8 |
| | | 6.1.1 Primary Efficacy Measures | 8 |
| | | 6.1.2 Secondary Efficacy Measure | 9 |
| | 6.2 | Other Efficacy Measure1 | 9 |
| | 6.3 | Safety Measure1 | 9 |
| | 6.4 | Other Measures1 | |
| 7 | Study | Materials1 | |
| | 7.1 | Study Drug(s)1 | |
| | | 7.1.1 Regimens | |
| | | 7.1.2 Dispensation Schedule | |
| | | 7.1.3 Instructions for Use | 9 |
| | 7.2 | Other Study Supplies2 | |
| 8 | Study | Methods and Procedures2 | |
| | 8.1 | Participant Entry Procedures2 | |
| | | 8.1.1 Overview | |
| | | 8.1.2 Informed Consent | |
| | | 8.1.3 Washout Intervals | |
| | | 8.1.4 Procedures for Final Study Entry | |
| | | 8.1.5 Methods for Assignment to Treatment Groups | |
| | 8.2 | Concurrent Therapies | |
| | | 8.2.1 Prohibited Medications/Treatments | |
| | | 8.2.2 Escape Medications | |
| | | 8.2.3 Special Diet or Activities | |
| | 8.3 | Examination Procedures | |
| | | 8.3.1 Procedures to be Performed at Each Study Visit with Regard to Stud | • |
| | | Objectives(s)2 | 8 |

| | 8.4 | Schedu | ale of Visits, Measurements and Dosing | 30 |
|---|---|---|---|---|
| | | 8.4.1 | Scheduled Visits | 30 |
| | | 8.4.2 | Unscheduled Visits | 30 |
| | 8.5 | Compl | iance with Protocol | 31 |
| | 8.6 | Subjec | t Disposition | 31 |
| | | 8.6.1 | Completed Subjects | 31 |
| | | 8.6.2 | Discontinued Subjects | 31 |
| | 8.7 | Study ' | Termination | 32 |
| | 8.8 | Study | Duration | 32 |
| | 8.9 | Monito | oring and Quality Assurance | 32 |
| 9 | safet | y definit | tions, safety monitoring and reporting | 32 |
| | 9.1 | Advers | se Event | 32 |
| | | 9.1.1 | Severity | 32 |
| | | 9.1.2 | Relationship to Study Drug | 33 |
| | | 9.1.3 | Expectedness | 33 |
| | 9.2 | Seriou | s Adverse Events | 34 |
| | 9.3 | Proced | lures for Reporting Adverse Events | 34 |
| | | 9.3.1 | Reporting a Suspected Unexpected Adverse Reaction | 35 |
| | | 9.3.2 | Reporting a Serious Adverse Event | 35 |
| | 9.4 | Proced | lures for Unmasking of Study Drug | 35 |
| | 9.5 | Type a | and Duration of the Follow-up of Subjects after Adverse Even | nts36 |
| 10 | Stati | | 1alysis | |
| | 10.1 | | e Size and Power Considerations | |
| | 10.2 | Analys | sis Populations | 36 |
| | | 10.2.1 | Intention-To-Treat Population | |
| | | 10.2.2 | Safety Population | |
| | 10.3 | | ical Hypotheses | |
| | 10.4 | | ical Analysis | |
| | | 10.4.1 | General Considerations | |
| | | 10.4.2 | Unit of Analysis | |
| | | 10.4.3 | Subject Demographics and Baseline Characteristics | |
| | | 10.4.4 | Primary Efficacy Analysis | |
| | | 10.4.5 | Secondary Efficacy Analysis | |
| | | 10.4.6 | Other Efficacy Analysis | |
| | | 10.4.7 | Safety Analysis | |
| | | 10.4.8 | Interim Analysis | 39 |
| 11 | | | with Good Clinical Practices, Ethical Considerations, and | |
| | | | ve Issues | |
| | 11.1 | | tion of Human Subjects | |
| | | 11.1.1 | Subject Informed Consent | |
| | | 11.1.2 | Institutional Review Board Approval | |
| | 11.2 | | l Conduct of Study | |
| | 11.3 | | t Confidentiality | |
| | 11.4 | Docum | nentation | 40 |


| | | 11.4.1 | Retention of Documentation | 40 |
|---|---|---|---|---|
| | 11.5 | Labeli | ng, Packaging, Storage, Accountability, and Return or Dis | posal of |
| | | Study | Drug | 41 |
| | | | Labeling/Packaging | |
| | | | Storage of Investigational Drug / Placebo | |
| | | | Accountability of Study Drug | |
| | | | Return or Disposal of Study Drug | |
| | 11.6 | | ding of Data on Source Documents and Electronic Case Re | |
| | | Forms | • | 41 |
| | 11.7 | Handli | ing of Biological Specimens | 42 |
| | 11.8 | | ations | |
| 12 | Refe | | | |
| 13 | | | | |
| App | | | dule of Visits and Measurements | |
| | | | nination Procedures, Tests, Equipment, and Techniques | |
| 11 | | | y Procedures | |
| | | | iomicroscopy | |
| | | - | orescein Staining | |
| | | | xamination | |
| | | | Test with Topical Anesthesia | |
| | | | ace Disease Index <sup>©</sup> | |
| | | | Score (EDS) Using a Visual Analog Scale (VAS) | |
| | | | Ocular Discomfort Scale | |
| App | | | sor Approvals | |
| | | | stigator's Signature | |
| 1. 1. | | | 0 0 | |

# LIST OF ABBREVIATIONS

| AE | Adverse event |
|-------------------|-------------------------------------------------------|
| ANCOVA | Analysis of covariance |
| BCVA | Best corrected visual acuity |
| BID | Two times a day |
| CAE® | Controlled adverse environment |
| CFR | Code of Federal Regulations |
| CI | Confidence interval |
| CRF | Case report form |
| EDS | Eye Dryness Score |
| DED | Dry eye disease |
| HIPAA | Health Information Portability and Accountability Act |
| IB | Investigator's Brochure |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| ITT | Intention to Treat |
| logMAR | Logarithm of the minimum angle of resolution |
| LS | Least Square |
| MAD | Mucosal Atomization Device |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple imputation |
| μL | microliter |
| mm | Millimeter |
| nAChR | Nicotinic acetylcholine receptor |
| OSDI <sup>©</sup> | Ocular Surface Disease Index <sup>©</sup> |
| PP | Per Protocol |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| TEAE | Treatment-emergent adverse event |
| US | United States |


# INTRODUCTION






#### 2 STUDY OBJECTIVES

The objective of this study is to evaluate the safety and effectiveness of OC-01 nasal spray compared to placebo on signs and symptoms of DED.

### 3 CLINICAL HYPOTHESES

This study is testing the hypothesis that OC-01 nasal spray is superior to placebo in treating the signs and symptoms of DED.


#### 4 OVERALL STUDY DESIGN

Protocol OPP-002 is a Phase 2, multicenter, randomized, double-masked, placebo-controlled study designed to evaluate the safety and efficacy of OC-01 nasal spray in adult participants with DED. Approximately 160 subjects at least 22 years of age with a physicians' diagnosis of dry eye disease and meeting all other study eligibility criteria will be randomized to receive an application of OC-01 or placebo twice daily (BID) for 4 weeks.

Participants who terminate early during the application period will be asked to complete safety assessments (if the participants agree) prior to study exit. Participants who are terminated early from the study will not be replaced.

#### 5 STUDY POPULATION

#### 5.1 Number of Subjects

Approximately 160 participants (approximately 40 per arm) will be enrolled at at least three sites in the US. Subjects will be randomized 1:1:1:1 to receive one of the following four dose assignments. All doses will be delivered as a 50 microliter (μL) intranasal spray in each nostril BID for a total of 6 weeks:

- Placebo (vehicle) [control]
- 0.02% OC-01 (varenicline tartrate) nasal spray [low dose]
- 0.1% OC-01 (varenicline tartrate) nasal spray [medium dose]
- 0.2% OC-01 (varenicline tartrate) nasal spray [high dose]

#### 5.2 Study Population Characteristics

All subjects must be at least 22 years of age, of either gender, and of any race, and must meet all inclusion criteria and none of the exclusion criteria.

#### 5.3 Inclusion Criteria

Subjects must:

2. Have used and/or desired to use an artificial tear substitute for dry eye symptoms within 6 months prior to Visit 1







6. Have had any intraocular surgery (such as cataract surgery), extraocular surgery (such as blepharoplasty) in either eye within three months or refractive surgery (e.g. laser epithelial keratomileusis, laser-assisted in-situ keratomileusis, photorefractive keratectomy or corneal implant) within twelve months of Visit 1



- 12. Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
- 13. Have a known hypersensitivity to any of the procedural agents or study drug components




17. Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject



investigational drug or device within 30 days prior to Visit 1

#### 5.5 Withdrawal Criteria

If at any time during the study the Investigator determines that a subject's safety has been compromised, the subject may be withdrawn from treatment, but will be followed for safety for the duration of the study, unless they refuse to attend follow-up visits.

Subjects may withdraw consent from the study at any time.

Sponsor and/or Investigator may discontinue any subject from study treatment for non-compliance or any valid medical reason during the course of the study (see Section 8.6.2).

#### 6 STUDY PARAMETERS

#### 6.1 Efficacy Measures

#### 6.1.1 Primary Efficacy Measure

The following primary endpoints will be tested:

• Schirmer's Test at Visit 5 (Day 28)


#### 6.1.2 Secondary Efficacy Measure

• EDS at Visit 4 (Day 21)

#### **6.2** Other Efficacy Measures

• Patient Reported Outcome: Ocular Discomfort Scale

• Corneal Staining

#### 6.3 Safety Measure

• Adverse Events

#### 6.4 Other Measures

• Urine pregnancy test (Visit 1 and Visit 4/ET)

#### 7 STUDY MATERIALS

#### 7.1 Study Drug(s)

#### 7.1.1 Regimens

The study drug will be delivered as a 50 microliter ( $\mu L$ ) intranasal spray in each nostril BID:

- Placebo (vehicle)
- 0.02% OC-01 (varenicline tartrate) [low dose]
- 0.1% OC-01 (varenicline tartrate) [medium dose]
- 0.2% OC-01 (varenicline tartrate [high dose]

#### 7.1.2 Dispensation Schedule

- At Visit 1, qualified subjects will be randomized and the first dose of study drug will be administered in office. The second daily administration will happen at home.
- At Visit 4 subjects will receive their first daily dose of study drug during CAE® exposure. The second daily administration will happen at home.
- At Visit 2, Visit 3, and Visit 5 the first daily dose of study drug will be administered in office concurrent with Schirmer's testing. The second daily administration will happen at home.
- Between clinic visits, subjects will self-administer OC-01 BID as a 50  $\mu$ L intranasal spray in each nostril.

#### 7.1.3 <u>Instructions for Use</u>





Figure 2






Figure 4


# Administration



Figure 5



Figure 6




Figure 7








Figure 10




Figure 11


### 7.2 Other Study Supplies

- Urine pregnancy test kits
- Fluorescein sodium solution or fluorescein strips
- Schirmer's test strips
- Proparacaine

#### 8 STUDY METHODS AND PROCEDURES

#### 8.1 Participant Entry Procedures

#### 8.1.1 Overview

Participants as defined by the criteria in Sections 5.2, 5.3, and 5.4 will be considered for entry into this study.

#### 8.1.2 Informed Consent

Prior to a participant's enrollment in the trial (i.e., prior to any study-related procedures), the study will be discussed with each potential participant and participants wishing to participate must be administered and provide written informed consent using an Institutional Review Board (IRB)-approved informed consent form (ICF). The ICF must be the most recent version that has received approval by a properly constituted IRB.

#### 8.1.3 Washout Intervals

Prohibited medications, treatments, and activities are outlined in the Exclusion Criteria (Section 5.4).

#### 8.1.4 Procedures for Final Study Entry

Subjects must meet all inclusion criteria and none of the exclusion criteria.

#### 8.1.5 Methods for Assignment to Treatment Groups

Each subject who enters the screening period for the study (defined as the point at which the subject signs the informed consent form (ICF) receives a unique subject identification number before any study-related activities/procedures are performed. This number will be used to identify the subject throughout the clinical study and must be used on all study documentation related to that subject.

The subject identification number must remain constant throughout the entire clinical study. This number will not necessarily be the same as the randomization number.

Subjects who meet the eligibility requirements will be randomly assigned to 1 of 4 treatment groups.


#### 8.2 Concurrent Therapies



#### 8.3 Examination Procedures

#### 8.3.1 Procedures to be Performed at Each Study Visit with Regard to Study Objectives(s)

The following procedures will be performed (see Appendix 2 for description).

#### Screening/Visit 1 (Day 1): Screening and Schirmer's Test Evaluation

- Informed consent/Health Information Portability and Accountability Act (HIPAA) consent
- Demographic data, medical history, prior medication (s), and ocular history
- Eligibility Criteria
- Urine pregnancy test (if applicable)
- OSDI<sup>©</sup> questionnaire
- EDS (visual analog scale)
- Ocular Discomfort Scale
- BCVA (pre-and post-treatment procedures)
- Slit lamp biomicroscopy (pre-and post-treatment procedures)
- Corneal fluorescein staining
- Schirmer's Test<sup>3</sup> (pre- and post- treatment procedures)
- Schirmer's Test with nasal stimulation (cotton swab)<sup>4</sup>
- Intranasal examination
- Randomization


<sup>&</sup>lt;sup>3</sup> Procedure will occur after corneal fluorescein staining

<sup>&</sup>lt;sup>4</sup> Schirmer's test with nasal stimulation will occur 10 minutes after the first Schirmer's test

- Dispense new study drug/placebo intranasal applicator
- Administration of study drug/placebo concurrently with Schirmer's Test

- Concomitant Medications
- AE Query

#### Visit 2 (Day 7 ±2): Schirmer's Test Evaluation

- BCVA (pre-and post-treatment)
- Slit lamp biomicroscopy (pre-and post-treatment)
- Administration of study drug/placebo
- Schirmer's Test (post-treatment)
- Concomitant Medications
- AE Query

#### Visit 3 (Day 14 ±2): Schirmer's Test Evaluation

- BCVA (pre-and post-treatment)
- Slit lamp biomicroscopy (pre-and post-treatment)
- Administration of study drug/placebo
- Schirmer's Test (concurrent with treatment)
- Dispense new study drug/placebo intranasal applicator
- Concomitant Medications
- AE Query

# Visit 4 (Day 21 ±2): CAE® Evaluation

#### **Pre- CAE® Procedures:**

- Urine pregnancy test (if applicable)
- EDS (visual analog scale)
- Ocular Discomfort Scale
- Concomitant Medications
- AE Query

#### **Pre-Treatment CAE® Evaluation**

- EDS (visual analog scale) until threshold is met
- Ora Calibra® Ocular Discomfort Scale until threshold is met

#### ADMINISTRATION OF INVESTIGATIONAL DRUG/PLACEBO

Treatment with Investigational drug/placebo will be administered upon a participant's reporting an Ocular Discomfort score  $\geq 3$  at two or more consecutive time points in at least one eye during CAE® exposure (participants with an Ocular Discomfort rating of 3


or 4 at time = 0 for an eye must report an Ocular Discomfort rating of 4 for two consecutive measurements for that eye) using the Scale. Participants will resume symptom assessments every 5 minutes starting 1 minute after the application ends.

#### **Post-Treatment CAE®** Evaluation

- EDS (visual analog scale)
- Ocular Discomfort Scale
- BCVA (at investigator's discretion as needed)
- Slit lamp biomicroscopy (at investigator's discretion as needed)
- AE Query

#### Visit 5 (Day 28 ±2): Schirmer's Test Evaluation

- BCVA (pre-and post-treatment)
- Slit lamp biomicroscopy (pre-and post-treatment)
- Intranasal examination
- Administration of study drug/placebo
- Schirmer's Test (concurrent with treatment)
- EDS (visual analog scale; post-treatment)
- Corneal fluorescein staining (post-treatment)
- Concomitant Medications
- AE Query

#### **Early Termination (if applicable)**

- BCVA
- Slit lamp biomicroscopy
- Intranasal examination
- Urine pregnancy test (if applicable)
- Concomitant Medications
- AE Query

# 8.4 Schedule of Visits, Measurements and Dosing

#### 8.4.1 Scheduled Visits

Refer to Appendix 1 for a schedule of visits and measurements.

#### 8.4.2 Unscheduled Visits

These visits may be performed in order to ensure subject safety. All procedures performed at an unscheduled visit will be recorded in the source documents and on the Unscheduled Visit


eCRF pages. Any procedure indicated in the eCRF that is not performed should be indicated as "Not done."

Evaluations that may be conducted at an Unscheduled Visit include:

- Slit-lamp Biomicroscopy;
- Visual Acuity;
- Intranasal Examination;
- Urine Pregnancy Test (if applicable);
- Assessment of AEs;
- Assessment of concurrent medications and/or treatments; and
- Any other assessments needed in the judgment of the investigator.

#### 8.5 Compliance with Protocol

Subjects will be instructed on the proper use and storage of the study drug at Visits 1, 2, 3, and 4, and provided with written instructions upon dispensation of their study drug at Visit 1 and Visit 3.

#### 8.6 Subject Disposition

#### 8.6.1 Completed Subjects

A completed subject is one who has completed 4 weeks of study visits.

#### 8.6.2 Discontinued Subjects

Subjects may be discontinued from treatment, or from involvement in the study at any time prior to their completion of the study due to:

- AEs:
- unmasking when medically necessary;
- protocol violations;
- administrative reasons (e.g., inability to continue, lost to follow-up);
- sponsor termination of study;
- subject choice (e.g. withdrawal of consent); and
- other

Note: In addition, any subject may be discontinued from treatment or from study involvement from any sound medical reason at the discretion of the investigator (after consultation with the Sponsor) or Sponsor.

Notification of a subject discontinuation and the reason for discontinuation will be made to Ora and/or Sponsor and will be clearly documented on the eCRF.

Discontinued subjects will not be replaced.


#### 8.7 Study Termination

The study may be stopped at any time by the Investigator and/or Ora after consultation with the Sponsor, with appropriate notification.

#### 8.8 Study Duration

An individual subject's participation will involve 5visits over approximately 4-weeks (28 days)

#### 8.9 Monitoring and Quality Assurance



# 9 SAFETY DEFINITIONS, SAFETY MONITORING AND REPORTING

#### 9.1 Adverse Event

An adverse event (AE) is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not the event is considered drug-related. An AE can therefore be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease occurring after the subject started dosing with the study drug, without any judgment about causality. Any pre-existing medical condition that worsens after administration of the study drug will also be considered a new AE.

Study drug includes the investigational drug under evaluation and placebo.

Documentation regarding the AE should be made as to the nature, date of onset, end date, severity, relationship to study drug, action(s) taken, seriousness, and outcome of any sign or symptom observed by the Investigator or reported by the subject upon indirect questioning.

#### 9.1.1 Severity

Severity of an AE is defined as a qualitative assessment of the degree of intensity of an AE as determined by the investigator or reported to him/her by the patient/subject. The assessment




of severity is made irrespective of relationship to study drug or seriousness of the event and should be evaluated according to the following scale:

- *Mild:* Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- *Moderate*: Event is bothersome, possibly requiring additional therapy, and may interfere with the subject's daily activities.
- Severe: Event is intolerable, necessitates additional therapy or alteration of therapy, and interferes with the subject's daily activities.

#### 9.1.2 Relationship to Study Drug

The relationship of each AE to the investigational product should be determined by the investigator (in a blinded manner) using these explanations:

- *Definite:* When there are good reason and sufficient documentation to demonstrate a direct causal relationship between investigational product and AE
- *Probable:* When there are good reasons and sufficient documentation to assume a causal relationship in the sense of plausible, conceivable, likely but not necessarily highly probable
- *Possible:* When there is sufficient information to accept the possibility of a causal relationship in the sense of not impossible and not unlikely, although the connection is uncertain or doubtful, for example; due to missing data or insufficient evidence.
- *None:* When there is sufficient information to accept a lack of a causal relationship, in the sense of impossible and improbable.
- *Unclassified:* When the causal relationship is not assessable for whatever reason due to insufficient evidence, conflicting data or poor documentation.

#### 9.1.3 Expectedness

The expectedness of an AE should be determined based upon existing safety information about the study drug using these explanations:

- *Unexpected:* An AE that is not listed in the Investigator's Brochure (IB) or is not listed at the specificity or severity that has been observed.
- Expected: An AE that is listed in the IB at the specificity and severity that has been observed.
- *Not Applicable:* Any AE that is unrelated to the study drug.

AEs that are mentioned in the IB as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug but are not specifically mentioned as occurring with the particular drug under investigation are to be considered unexpected.

The investigator should initially classify the expectedness of an AE, but the final classification is subject to the Medical Monitor's determination.


#### 9.2 Serious Adverse Events

An AE is considered "serious" (SAE) if, in the view of either the investigator or Sponsor, it results in any of the following outcomes:

- Death
- A life-threatening AE

Note: An AE is considered "life-threatening" if, in the view of either the investigator or Sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an AE that, had it occurred in a more severe form, might have caused death.

• Inpatient hospitalization or prolongation of existing hospitalization

Note: The term "inpatient hospitalization" refers to any inpatient admission (even if less than 24 hours). For chronic or long-term inpatients, inpatient admission includes transfer within the hospital to an acute/intensive care inpatient unit. Inpatient hospitalization does not include: emergency room visits; outpatient/same-day/ambulatory procedures; observation/short stay units; rehabilitation facilities; hospice facilities; nursing homes; or clinical research/phase 1 units.

Note: The term "prolongation of existing hospitalization" refers to any extension of an inpatient hospitalization beyond the stay anticipated or required for the reason for the initial admission as determined by the investigator or treating physician.

• A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions

Note: An SAE specifically related to visual threat would be interpreted as any potential impairment or damage to the subject's eyes (e.g., hemorrhage, retinal detachment, central corneal ulcer or damage to the optic nerve).

• A congenital anomaly/birth defect in an offspring of a study subject.

Important medical events that may not result in death, are life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

#### 9.3 Procedures for Reporting Adverse Events

All AEs and their outcomes must be reported to Ora, the Sponsor, and the IRB/IEC as required by the IRB/IEC, federal, state, or local regulations and governing health authorities and recorded on the appropriate eCRF.


#### 9.3.1 Reporting a Suspected Unexpected Adverse Reaction

All AEs that are 'suspected' and 'unexpected' are to be reported to Ora, the Sponsor and the IRB/IEC as required by the IRB/IEC, federal, state, or local regulations and governing health authorities.

#### 9.3.2 Reporting a Serious Adverse Event

To ensure subject safety, all SAEs, regardless of relationship to the study drug, must be immediately reported. All information relevant to the SAE must be recorded on the appropriate CRFs. The investigator is obligated to pursue and obtain information requested by Ora and/or the Sponsor in addition to that information reported on the CRF. All subjects experiencing a SAE must be followed up and the outcome reported.

In the event of a SAE, the investigator must notify Ora and the Sponsor immediately; obtain and maintain in his/her files all pertinent medical records, information, and medical judgments from colleagues who assisted in the treatment and follow-up of the subject; provide Ora and the Sponsor with a complete case history, which includes a statement as to whether the event was or was not suspected to be related to the use of the study drug; and inform the IRB of the SAE within their guidelines for reporting SAEs.

Contact information for reporting SAEs:



# 9.4 Procedures for Unmasking of Study Drug

All subjects, investigators, and study personnel involved with the conduct of the study will be masked with regard to treatment assignments. When medically necessary, the investigator may need to determine what treatment regimen has been assigned to a subject. When possible (i.e., in non-emergent situations), Ora and/or the Sponsor should be notified before unmasking study drug. The unmasked subject will continue the study if warranted by the Investigator in consultation with the Medical Monitor.


# 9.5 Type and Duration of the Follow-up of Subjects after Adverse Events

Sponsor: Oyster Point Pharma, Inc

The investigator will follow unresolved AEs to resolution until the subject is lost to follow-up or until the AE is otherwise classified. Resolution means the subject has returned to baseline state of health or the Investigator does not expect any further improvement or worsening of the AE. If the patient is lost to follow-up, the Investigator should make 3 reasonable attempts to contact the patient via telephone, post, or certified mail. All follow-up will be documented in the subject's source document. Non-serious AEs identified on the last scheduled contact must be recorded on the AE eCRF with the status noted.

If the Investigator becomes aware of any new information regarding an existing SAE (i.e., resolution, change in condition, or new treatment), a new SAE/Unanticipated Report Form must be completed and faxed to Ora within 24 hours of the site's awareness of the new information. The original SAE form is not to be altered. The report should describe whether the event has resolved or continues and how the event was treated.

#### 10 STATISTICAL ANALYSIS

Statistical considerations and methods of analyses for this study are provided below; the accompanying Statistical Analysis Plan (SAP) contains complete details of the planned analyses.

#### 10.1 Sample Size and Power Considerations

The study will randomize approximately 160 subjects in a 1:1:1:1 ratio to the four treatment groups. Approximately 38 subjects in each treatment group are expected to complete their assigned treatment and have endpoint assessments at Visit 5.

The primary efficacy endpoint is change in Schirmer's Test Score (STS) from baseline to Visit 5. Two-sided t-tests at a Dunnett-corrected 5% significance level will be used.

A previous Phase 2a study (OCUP-001) showed a standard deviation (SD) of approximately 10 units for change in STS. Assuming a standard deviation of 10 units and a mean difference of 6 units between the high or medium doses of OC-01 and placebo, the probability (i.e., the power) that at least one of the two comparisons would be significant is roughly 80%.

#### **10.2** Analysis Populations

#### 10.2.1 Intention-To-Treat Population

The intent-to-treat (ITT) population will include all randomized subjects. Analyses using the ITT population will group subjects according to the treatment to which they were randomized.


### 10.2.2 Safety Population

The safety population will include all randomized subjects who received at least one dose of the study drug. Analysis on the safety population will group subjects according to the treatment actually received.

### 10.3 Statistical Hypotheses

The mean change in STS from baseline to Visit 5 is denoted as  $\mu_p$ ,  $\mu_l$ ,  $\mu_m$ , and  $\mu_h$  for placebo, OC-01 low dose, OC-01 medium dose, and OC-01 high dose, respectively.

Ho1: 
$$\mu_p = \mu_m = \mu_h$$

$$H_{11}$$
:  $\mu_p \neq \mu_m$ , or  $\mu_p \neq \mu_h$ 

No hypothesis is made comparing the OC-01 low dose group to placebo. A successful outcome will be one that rejects the null hypothesis for a given dose.

### 10.4 Statistical Analysis




### 10.4.3 Subject Demographics and Baseline Characteristics

Continuous summary statistics will be generated for age in years by treatment group and for all subjects. Discrete summary statistics will be generated for the following qualitative demographic variables: age category, gender, ethnicity, race, and other baseline intranasal examination results, tabulated by treatment group and for all subjects. Individual subject data listings will support the Summary tables.

### 10.4.4 Primary Efficacy Analysis



### 10.4.7 Safety Analysis

All safety analyses will be performed on the safety population.


The safety of OC-01 will be assessed primarily by the incidence of AEs. An AE will be considered a treatment-emergent AE (TEAE) if it occurs or worsens on or after initiation of treatment. An overall summary of TEAEs will be presented including the number of events and the number of subjects with events (along with percentages) by treatment group for TEAEs in several categories base on seriousness, relationship to treatment, and severity.

Other safety endpoints including visual acuity, slit-lamp biomicroscopy and intranasal examination will be summarized by treatment group and visit using descriptive statistics. Changes or shifts from baseline will be summarized where appropriate. For assessments performed by eye, study eye and fellow eye will be summarized separately. In addition, shifts from baseline to worst on-treatment value for ocular safety assessments will be summarized.

The SAP will present methods of analysis of these defined parameters in detail.

### 10.4.8 Interim Analysis

No interim analysis planned for this study.

# 11 COMPLIANCE WITH GOOD CLINICAL PRACTICES, ETHICAL CONSIDERATIONS, AND ADMINISTRATIVE ISSUES

This study will be conducted in compliance with the protocol, Good Clinical Practices, including the International Conference on Harmonization (ICH) Guidelines, and in general, consistent with the Declaration of Helsinki. In addition, all applicable local, state, and federal requirements relevant to the use of study drugs in the countries involved will be adhered to.

### 11.1 Protection of Human Subjects

### 11.1.1 Subject Informed Consent

Informed consent/assent must take place before any study specific procedures are initiated. Signed and dated written informed consent must be obtained from each subject and/or from the subject's parent or legal guardian prior to enrollment into the study. If the subject is under the legal age of consent, the consent form must be signed by a legal guardian or as required by state and/or local laws and regulations.

All informed consent/assent forms must be approved for use by the Sponsor and receive approval/favorable opinion from an IRB prior to their use. If the consent form requires revision (e.g., due to a protocol amendment or significant new safety information), it is the investigator's responsibility to ensure that the amended informed consent is reviewed and approved by Ora prior to submission to the governing IRB and that it is read, signed and dated by all subjects subsequently enrolled in the study as well as those currently enrolled in the study.

If informed consent is taken under special circumstances (oral informed consent), then the procedures to be followed must be determined by Ora and/or Sponsor and provided in writing by Ora and/or Sponsor prior to the consent process.


### 11.1.2 Institutional Review Board Approval

This study is to be conducted in accordance with IRB regulations [U.S. 21 Code of Federal regulations (CFR) Part 56.103]. The investigator must obtain appropriate IRB approval before initiating the study and re-approval at least annually.

Only an IRB-approved version of the informed consent form will be used.

### 11.2 Ethical Conduct of Study

This study will be conducted in accordance with the ethical principles that originated with the Declaration of Helsinki.

### 11.3 Subject Confidentiality

All personal study subject data collected and processed for the purposes of this study should be maintained by the investigator and his/her staff with adequate precautions as to ensure that the confidentiality of the data in accordance with local, state, and federal laws and regulations.

Monitors, auditors and other authorized representatives of Ora, the Sponsor, the IRB approving this study, the Food and Drug Administration, the Department of Health and Human Services, other domestic government agencies, and other foreign regulatory agencies will be granted direct access to the study subject's original medical and study records for verification of the data and/or clinical trial procedures. Access to this information will be permitted to the aforementioned individuals to the extent permitted by law.

A report of the results of this study may be published or sent to the appropriate health authorities in any country in which the study drug may ultimately be marketed, but the subject's identity will not be disclosed in these documents.

### 11.4 Documentation

Source documents may include a subject's medical records, hospital charts, clinic charts, the investigator's study subject files, as well as the results of diagnostic tests such as X-rays, laboratory tests, and electrocardiograms. The investigator's copy of the CRFs serves as the investigator's record of a subject's study-related data.

### 11.4.1 Retention of Documentation

All study related correspondence, subject records, consent forms, record of the distribution and use of all study drug and copies of CRFs should be maintained on file for at least two years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region; or until at least two years have elapsed since the formal discontinuation of clinical development of the study drug. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the Sponsor. It is the responsibility of the


Sponsor to inform the investigator/institution as to when these documents no longer need to be retained.

If the responsible investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian.

# 11.5 Labeling, Packaging, Storage, Accountability, and Return or Disposal of Study Drug

### 11.5.1 <u>Labeling/Packaging</u>

Investigational drug will be provided in multi-use intranasal applicator that will be assigned at randomization for use during the first 14 days of study. A second multi-use intranasal applicator will be provided at Visit 3 (Day 14) for use during days 14-28.

### 11.5.2 Storage of Investigational Drug / Placebo

The investigational drug / placebo must be stored in a secure area accessible only to the investigator and his/her designee(s). Study drug(s) must be refrigerated (2-8°C, Do Not Freeze), protected from light, and secured at the investigational site in a locked container.

### 11.5.3 Accountability of Study Drug

The investigational drug / placebo is only prescribed by the principal investigator or his/her named sub investigator(s), and is to only be used in accordance with this protocol. The study drugs must only be distributed to subjects properly qualified under this protocol to receive study drug. The investigator must keep an accurate accounting of the study drugs by maintaining a detailed inventory. This includes the amount of study drugs received by the site, amount dispensed to subjects, amount returned to the site by the subjects, and the amount returned to the Sponsor upon the completion of the study.

### 11.5.4 Return or Disposal of Study Drug

All study drugs will be returned to the Sponsor or their designee for destruction.

# 11.6 Recording of Data on Source Documents and Electronic Case Reports Forms

All subject data will be captured in the subject source documents which will be transcribed in the eCRFs. The investigator is responsible for ensuring that study data is completely and accurately recorded on each subject's eCRF, source documents, and all study-related materials. All study data should also be attributable, legible, contemporaneous, and original. Recorded datum should only be corrected in a manner that does not obliterate, destroy, or render illegible the previous entry (e.g., by drawing a single line through the incorrect entry and writing the revision next to the corrected data). An individual who has corrected a data


entry should make clear who made the correction and when, by adding to the correction his/her initials as well as the date of the correction.

Data entry of all enrolled and randomized subjects will use software that conforms to 21 CFR Part 11 requirements, and will be performed only by staff who have been trained on the system and have access to the system. Data will not be entered for screen failure subjects. An audit trail will be maintained within the electronic system to capture all changes made within the eCRF database. After the end of the study and database lock, electronic copies of all applicable subjects' eCRFs will be provided to each Investigator Site to be maintained on file by the Investigator.

### 11.7 Handling of Biological Specimens

Not applicable.

### 11.8 Publications

The study will be documented in a final report, which will contain appropriate statistical analysis and medical overview. No individual site or Investigator may publish or present any results from the study until the Sponsor completes a joint, multi-center publication of the trial results is made by Sponsor in conjunction with various participating Investigators and appropriate sites contributing data and comments. Subsequently, individual Investigators may request to publish or present results from the trial; however, approval will be at the sole discretion of the Sponsor. Should the foregoing language be in conflict with the language addressing publication in the clinical trial agreement, the language in the Clinical Trial Agreement will prevail.


### 12 REFERENCES










# 13 APPENDICES

CONFIDENTIAL

# APPENDIX 1: SCHEDULE OF VISITS AND MEASUREMENTS

| ALLENDIA I. SCHEDOLE OF VISITS AND MEASONEMENTS | | | CITCIA | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screen/<br>Visit 1 | | Visit 2 | | Visit 3 | | Visit 4<br>(Day 21 ±2) | it 4<br>:1 ±2) | | Visit 5 | |
| Procedure | Day 1 | Days<br>2-6 | Day 7 ±2 | Days<br>8-13 | Day 14 ±2 | Days<br>15-20 | Pre-CAE® | Post-CAE® | Days<br>22-27 | Day 28 ±2 | ET |
| Informed consent/HIPAA | × | | | | | | | | | | |
| Demographics | X | | | | | | | | | | |
| Medical history, prior medication(s), ocular history and updates | X | | | | | | | | | | |
| Eligibility criteria | X | | | | | | | | | | |
| Urine pregnancy test | X <sub>4</sub> | | | | | | X4 | | | | X <sub>4</sub> |
| OSDI® questionnaire | X | | | 3 | | | | | | | |
| Eye Dryness Score (EDS) | X | | | | | | X | Xs | | $X_2$ | |
| Ocular Discomfort Scale | × | | | | | | X | Xs | | | |
| BCVA | $X_1$ | | $^{1}X$ | | $X_1$ | | | X <sub>6</sub> | | $X_1$ | X |
| Slit lamp biomicroscopy | $X_1$ | | $X_1$ | 3 | $X_1$ | | | X <sub>6</sub> | | Xı | X |
| Corneal fluorescein staining | X | | | | | | | | | $X_2$ | |
| Schirmer's test | $X_1$ | | X | | X | | | | | X | |
| Schirmer's test with cotton swab stimulation | X | | | | | | | | | | |
| Intranasal examination | $X_1$ | | | | | | | | | X | X |
| Randomization | X | | | | | | | | | | |
| Administer investigational drug / placebo | X3 | X | $X_3$ | X | X3 | Х | Х | | Х | $X_3$ | |
| Dispense investigational drug / placebo | X | | | | X | | | | | | |
| Concomitant medications | X | | X | | X | | X | | | X | X |
| AE Query | X | | X | | X | | X | X | | X | X |
| | 1 | Over the second second second second | The second secon | Control of the last of the las | CONTRACTOR OF THE PROPERTY OF THE PARTY OF T | | The state of the s | THE CONTRACTOR OF THE PARTY OF | The second secon | | |

X<sub>1</sub> = Pre- and Post-treatment procedures; X<sub>2</sub> = Post-treatment procedures X<sub>3</sub> = Concurrent with Schirmer's Test; X<sub>4</sub> = For females of childbearing potential; X<sub>5</sub> = Procedure started at time 0 and then conducted every 5 minutes thereafter during the 120 minute CAE\* exposure; Xo = Procedure may be performed after CAE® exit at the Investigator's discretion as needed

# APPENDIX 2: EXAMINATION PROCEDURES, TESTS, EQUIPMENT, AND TECHNIQUES

Sponsor: Oyster Point Pharma, Inc.

The following examination procedures, tests, equipment and techniques are listed in this Appendix:

### **Visual Acuity Procedures**

LogMAR visual acuity must be assessed using an ETDRS chart. The procedure used will be consistent with the recommendations provided for using the ETDRS eye chart. Visual acuity should be evaluated at the beginning of each visit in the study (i.e., prior to slit lamp examination). Participants should use the most recent correction to attain their corrected distance visual acuity (CDVA); if they forget their spectacles, this prescription can be placed in a trial frame.

### Equipment

The visual acuity chart to be used is the ETDRS chart. If smaller reproduction (18" by 18", e.g., from Prevent Blindness) wall charts are used, the participant viewing distance should be exactly 10 feet (or as specified by the manufacturer). In ALL cases, for purposes of standardizing the testing conditions during the study, all sites must use only ETDRS Series 2000 Chart 1 & 2, and the right eye should be tested first. For reflectance (wall) charts, the chart should be placed frontally and be well illuminated.

### Measurement Technique

The chart should be at a comfortable viewing angle. The right eye should be tested first. The participant should attempt to read each letter, line-by-line, left to right, beginning with line 1 at the top of the chart. The participant should be told that the chart has letters only, no numbers. If the participant reads a number, s/he should be reminded that the chart contains no numbers, and the examiner should then request a letter in lieu of the number. The participant should be asked to read slowly, so as to achieve the best identification of each letter. S/he is not to proceed to the next letter until s/he has given a definite response.

If the participant changes a response (e.g., 'that was a "C" not an "O"') before s/he has read aloud the next letter, then the change must be accepted. If the participant changes a response having read the next letter, then the change is not accepted. The examiner should never point to the chart or to specific letters on the chart during the test.

A maximum effort should be made to identify each letter on the chart. When the participant says s/he cannot read a letter, s/he should be encouraged to guess. If the participant identifies a letter as one of two letters, s/he should be asked to choose one letter and, if necessary, to guess. When it becomes evident that no further meaningful readings can be made, despite encouragement to read or guess, the examiner should stop the test for that eye. However, all letters on the last line should be attempted as letter difficulties vary and the last may be the only one read correctly. The number of letters missed or read incorrectly should be noted.


### LogMAR Visual Acuity Calculations

The last line in which a letter is read correctly will be taken as the base logMAR reading. To this value will be added the number "N x 0.02" where 'N' represents the total number of letters missed up to and including the last line read. This total sum represents the logMAR visual acuity for that eye.

Example: Participant correctly reads 4 of 5 letters on the 0.2 line, and 2 of 5 letters on the 0.1 line.

| Base logMAR | = 0.1 |
|---|---|
| N (total number of letters incorrect on line 0.2 as well as 0.1) | = 4 |
| N x T (T=0.02) | = 0.08 |
| Base logMAR + (N x T) | = 0.1 + 0.08 |
| logMAR visual acuity | = 0.18 |

Repeat the procedure for the left eye.

In order to provide standardized and well-controlled assessments of visual acuity during the study, all visual acuity assessments at a single site must be consistently done using the same lighting conditions and same correction if possible during the entire study. If the same correction cannot be used (i.e., a participant broke his/her glasses), the reason for the change in correction should be documented.

Note: A clinically significant visual acuity decrease (defined as an increase of 0.22 or greater in logMAR score) from the Screening Visit (Visit 1) should be evaluated by the Investigator as a potential AE.


### Slit Lamp Biomicroscopy

Slit lamp biomicroscopy will be performed during the study. Observations will be graded as *Normal* or *Abnormal*. Abnormal findings, which are clinically significant, will be described.

Sponsor: Oyster Point Pharma, Inc.

### **Corneal Fluorescein Staining**

The examiner should instill 5  $\mu$ L of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. Alternatively, corneal staining can be assessed using 1.0 mg sodium fluorescein strips. After moistening the tip of the strip with sterile buffered saline, the excess is shaken into a waste bin with a sharp flick. The lower lid is then pulled down and the flat end of the tip should be gently applied to the inferior tarsal conjunctiva with the intent of not inducing reflex tearing and instilling a very small volume of dye.

The participant will be instructed to blink naturally several times without forced closure of the eyelid to distribute the fluorescein. In order to achieve maximum fluorescence, the examiner should wait at least two minutes after instillation before evaluating corneal fluorescein staining. A Wratten #12 yellow filter will be used to enhance the ability to grade fluorescein staining. The staining will be graded with the NEI Scale. The upper eyelid is lifted slightly to grade the entire corneal surface.




### **Intranasal Examination**

Qualified participants for the study must undergo an intranasal exam to make the final eligibility determination (e.g. severe nasal airway obstruction such as, severe septal deviation or inferior turbinate hypertrophy, or vascularized polyp seen on examination are reasons for exclusion). To monitor nasal mucosal integrity during the study for participant safety, an examination of the nasal cavities via an intranasal exam will be performed at the Screening Visit (after all other screening procedures have been completed). This examination will be performed by an Ear Nose and Throat (ENT) specialist, otolaryngologist or other suitably qualified medical practitioner (i.e. one who has been trained to perform intranasal exam). Still images or video may be captured. The procedure used for the intranasal exam can be conducted either by endoscopic examination or nasal specula.


### Schirmer's Test with Topical Anesthesia

At the Screening Visit, one basal Schirmer's test will be performed followed by a Schirmer's test with cotton swab nasal stimulation. The Schirmer's test with topical anesthetic will be used to assess tear production using the following steps:

Sponsor: Oyster Point Pharma, Inc.

- 1. Topical anesthetic drops such as 0.5% proparacaine hydrochloride or equivalent should be instilled in both eyes of the participant.
- 2. The participant will be instructed to keep the eyes gently closed for one minute.
- 3. After opening the eyes and allowing the eyes to recover for approximately one additional minute, excess moisture in the inferior fornix is gently removed with a spear.
- 4. Schirmer's strips (35 mm x 5 mm size filter paper strip) will be placed in each eye at the junction of the middle and lateral thirds of the lower eye lid.
- 5. Under ambient light, the participant will be instructed to look forward and to blink normally during the course of the test. The test should be performed in a room with no direct air on the participant's face.
- 6. The Schirmer's strips should remain in place until five minutes have elapsed or both strips have reached maximum score.
- 7. After five minutes, strips will be removed from both eyes and the amount of wetting will be recorded. The strips should be taped to the CRF.

### Schirmer's test using cotton swab nasal stimulation

At the Screening Visit, the Schirmer's test should be performed using cotton swab nasal stimulation. New anesthetic drops should be instilled following the same procedure specified in steps #1 to 3 above.

- 1. With new strips in place, the examiner should insert cotton swabs in the participant's two nostrils simultaneously and gently probe both nasal middle turbinates for approximately 30 seconds. After this, the examiner can simply hold the swabs in place, applying gentle pressure, and repeat probing intermittently as necessary.
- 2. Alternatively, the participant can be instructed to hold the cotton swabs and gently probe both nasal turbinates simultaneously, resting intermittently before probing again. The examiner should continuously coach the participant on how to perform this test properly.
- 3. The Schirmer's strips should remain in place until five minutes have elapsed or both strips have reached maximum score.

Both Schirmer's scores will be recorded and verified that they meet the inclusion criteria.







The EDS is an instrument that has been used in other


Chinical Trial Protocol #OPP-002


### APPENDIX 3: SPONSOR AND APPROVALS

Protocol Title: Multicenter, Randomized, Controlled, Double-Masked Clinical

Trial to Evaluate the Efficacy of OC-01 Nasal Spray on Signs and

Symptoms of Dry Eye Disease




### **APPENDIX 4: INVESTIGATOR'S SIGNATURE**

| <b>Protocol Title:</b> | Multicenter, Randomized, Control<br>Trial to Evaluate the Efficacy of O<br>Symptoms of Dry Eye Disease | |
|---|---|---|
| <b>Protocol Number:</b> | OPP-002 | |
| protocol, good clinical pall information supplied submitted to an Institution designation that the manager of the submitted to a designation that the manager of the supplies that the manager of the supplies that the manager of the supplies that the manager of the supplies that the manager of the supplies that the sup | d conduct the study diligently and in tractices and all applicable laws and by and the Sponsor in confident and Review Board (IRB) or another aterial is confidential. | regulations. I agree to maintain ace and, when this information is group, it will be submitted with |
| Signed: | | Date: |
| Name: | | <del>-</del> |
| Title: | | - |
| Site: | | - |
| Address: | | - |
| Phone Number: | | - |

